CLINICAL TRIAL: NCT00538291
Title: CA225103: A Phase II Study of a Combination of Cetuximab and Capecitabine in Patients With Metastatic Colorectal Cancer After Progression on Previous Fluoropyrimidine Containing Therapy
Brief Title: Cetuximab and Capecitabine in Treating Patients With Metastatic Colorectal Cancer That Failed Irinotecan Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to lack of efficacy.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05033; P30CA033572 (NIH); CHNMC-05033; CDR0000567432 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry

ARMS (1):
- Arm 1 (Experimental): Cetuximab 400mg/m2 IV on day 1 over 2 hours then 250 mg/m2 over 1 hour weekly + Xeloda(Capecitabine) 1000mg/m2 BID on days 1-14 repeated every 21 days.
  Interventions: Biological: cetuximab; Drug: capecitabine; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: polymorphism analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: immunohistochemistry staining method

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymorphism analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with capecitabine work in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic colorectal cancer treated with cetuximab and capecitabine that progressed on prior fluoropyrimidine-containing therapy comprising irinotecan with or without oxaliplatin.

Secondary

* To determine the progression-free survival and overall survival of patients treated with this regimen.
* To determine the tolerance to therapy in these patients.
* To assess biological correlates of response in available tissue biopsies and blood samples.

OUTLINE: Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood collection periodically for correlative studies. Samples are analyzed for expression of genes correlated with fluoropyrimidine responsiveness via quantitation RT-PCR; degree of expression of EGFR via immunohistochemistry; and expression pattern analysis via gene expression profiling and polymorphism.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal cancer
* Measurable disease
* Disease progression during prior fluoropyrimidine-containing therapy comprising irinotecan with or without oxaliplatin

  * Received standard first- and second-line irinotecan and oxaliplatin-based therapy

    * Patients who completed 1 prior treatment for metastatic disease but refused standard second-line therapy are eligible
  * Patients who's disease progressed within 6 months of previous therapy are eligible
* EGFR negative patients allowed
* No untreated or uncontrolled brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* ALT ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Serum creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No serious intercurrent infections or medical problems
* No active or uncontrolled infections
* No significant history of uncontrolled cardiac disease, including any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* No prior severe infusion reaction to a monoclonal antibody
* No known dihydropyrimidine dehydrogenase deficiency or evidence of past hypersensitivity to fluoropyrimidine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 2 prior treatments for metastatic colorectal cancer
* More than 2 weeks since prior therapy
* Prior radiotherapy allowed if < 30% of bone marrow involvement
* No other concurrent investigational agents
* No concurrent highly active antiretroviral therapy for HIV-positive patients
* No prior therapy that specifically and directly targets the EGFR pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 13
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 61 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by spiral CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Assessment after every 2 cycles of treatment, up to 1 year.
Population: The three patients not completing at least two courses of treatment were considered treatment failures and were included in efficacy analysis.
Measure: Number; unit: number of responding participants
Arm/Group | Arm 1
Number analyzed (Participants) | 13
number of responding participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of of 17 months.
Description: "Other" adverse events include all grades and attribution to treatment that are not included in "Serious" adverse events
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=13)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (23)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (5)
Fatigue (General disorders) | 12 (42)
Fever (General disorders) | 3 (3)
Injection site reaction (General disorders) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (20)
Alkaline phosphatase increased (Investigations) | 9 (20)
Aspartate aminotransferase increased (Investigations) | 11 (37)
Bilirubin increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 2 (2)
Hyperbilirubinemia (Investigations) | 2 (5)
Leukocyte count decreased (Investigations) | 5 (8)
Leukopenia (Investigations) | 1 (2)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Lymphopenia (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 3 (16)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (11)
Hypokalemia (Metabolism and nutrition disorders) | 1 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (11)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (9)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (7)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (7)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Ureteric hemorrhage (Renal and urinary disorders) | 2 (3)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 4 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 8 (15)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (16)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to a lack of efficacy (less than 2 of 13 patients responded to treatment in the first stage of a Simon's two stage design).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes